CLINICAL TRIAL: NCT06334874
Title: Study of the Efficacy and Safety of Astaxanthin as an Adjuvant Therapy for Community Acquired Pneumonia Patients.
Brief Title: Study of the Efficacy and Safety of Antioxidants Astaxanthin as an Adjuvant Therapy for Community Acquired Pneumonia Patients.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Fatma Makram Youssef, teaching assistant, pharmacy practice & clinical pharmacy department, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-FPFUE-32/2023
Record Dates: First submitted 2024-03-02; First posted 2024-03-28 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Active Comparator)
  Interventions: Drug: Astaxanthin Oral Capsule
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Astaxanthin Oral Capsule — 12 mg of astaxanthin oral capsule
  Arms: intervention
Drug: Placebo — starch placebo capsule
  Arms: placebo

SUMMARY:
Community acquired pneumonia (CAP) is one of the most common and morbid conditions encountered in clinical practice, which causes serious morbidity worldwide. In CAP, oxidative stress is linked to inflammation, demonstrated by increased production of interleukin (IL)-6 and tumor necrosis factor (TNF)-α, which attract inflammatory cells and increase oxidant production by these cells. Attenuation of oxidative stress via antioxidants would be expected to result in reduced pulmonary damage. Antioxidants have been found to be effective in alleviating lung injury and protecting against damage of other organs.

DETAILED DESCRIPTION:
The study will be randomized controlled trial, that will be carried out at ICU at El Matarya Teaching Hospital.

Prior to participation in the study, written informed consent will be obtained from the patients or their family.

Patients with the following criteria will be enrolled: age ≥ 18 year, having clinical symptoms suggestive of CAP such as cough (with or without sputum), fever (> 38.5°C), pleuritic chest pain or dyspnea and consolidations on computed Tomography (CT). Patients will be excluded from the study if having one of the following criteria: advanced age (≥70 years old), presence of severe immunosuppression (HIV infection, use of immune suppressants), malignancy, other concurrent infections, obstruction pneumonia (e.g., because of lung cancer), pneumonia developed within two weeks after hospital discharge, use of ASX before study entry, hypersensitivity to ASX, taking warfarin, taking other antioxidants such as vitamin C, vitamin E, glutathione, granulocytopenia (<1000 neutrophils/mm3), renal failure, liver failure, pregnant and lactating women, hemodynamically unstable patients.

Eligible CAP patients at El Matarya Teaching Hospital will be randomly assigned to either ASX group or control group. The ASX group will receive ASX (12mg/d) orally or enterally in addition to conventional therapy for CAP. [1,2] The control group will receive placebo orally or enterally in addition to conventional therapy for CAP. [2] The treatment duration will be from hospital admission till time of discharge for each CAP patient.

All patients will be subjected to the following:

A. Patient Data Collection:

1. Baseline characteristics: demographic data of the participants including: age, gender, weight, height, and body mass index (BMI).
2. Medication History: complete history of medication will be recorded for each patient including medications for comorbidities and past medication history as well as concomitant medications.
3. Medical History: patient history will be recorded including history of present illness as well as comorbidities.

B. Clinical Assessment:

1. Physical Examination: daily records of ABGS, body temperature, pulse, blood pressure, and respiratory rate will be collected, baseline and final readings will be used for analysis.
2. Biochemical Investigations:

2.1 The biochemical parameters include complete blood count with differential counts of total leukocyte count, lymphocytic count, liver function, renal functions, albumin level, creatinine level, alkaline phosphatase level, ferritin level, C-reactive protein, Prothrombin time (PT), activated partial thromboplastin time APTT, lipid profile and blood sugar level , baseline and final readings will be used for analysis.

2.2 Cytokine storm parameters (interleukin-6, tumor necrosis factor-α, and interleukin10) will be assessed at baseline and at the end of the study.

C. Severity Assessment: CURB-65 severity score that has been validated for predicting mortality of CAP, will be assessed at baseline and at the end of the study.[3] D. Radiological Assessment of CAP: computed tomography will be carried out before enrollment to confirm pneumonia diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Clinical: Having symptoms suggestive of CAP such as cough (with or without sputum), fever (> 38.5°C), pleuritic chest pain or dyspnea.
* Radiologic: consolidations on computed Tomography (CT).

Exclusion Criteria:

* Advanced age (≥70 years old). Presence of severe immunosuppression (HIV infection, use of immune suppressants).

Malignancy. Other concurrent infections, obstruction pneumonia (e.g., because of lung cancer).

Pneumonia developed within two weeks after hospital discharge. Use of ASX before study entry. Hypersensitivity to ASX. Taking warfarin.

* Taking other antioxidants such as vitamin C, vitamin E, glutathione.
* Granulocytopenia (<1000 neutrophils/mm3).
* Renal failure.
* Liver failure.
* Pregnant and lactating women.
* Hemodynamically unstable patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
change in IL-6 after treatment in the ASX group compared with those in the control group. | from time of randomization till seven days
  The primary endpoint indicators is the change in IL-6 after treatment in the ASX group compared with those in the control group.
change in IL-10 after treatment in the ASX group compared with those in the control group. | from time of randomization till seven days
  the primary endpoint indicators is the change in IL-10 after treatment in the ASX group compared with those in the control group.
change in tumor necrosis alpha after treatment in the ASX group compared with those in the control group. | from time of randomization till seven days
  the primary endpoint indicators is the change in tumor necrosis alpha after treatment in the ASX group compared with those in the control group.

SECONDARY OUTCOMES:
difference in CURB 65 scores after treatment in the ASX group compared with the control group. | from time of randomization till seven days
  CURB-65, also known as the CURB criteria, is a clinical prediction rule that has been validated for predicting mortality in pneumonia.
  The score is an acronym for each of the risk factors measured. Each risk factor scores one point, for a maximum score of 5:
  Confusion of new onset (defined as an AMTS of 8 or less) Blood Urea nitrogen greater than 7 mmol/L (19 mg/dL) Respiratory rate of 30 breaths per minute or greater Blood pressure less than 90 mmHg systolic or diastolic blood pressure 60 mmHg or less Age 65 or older
o Adverse drug reactions related to ASX as increase bowel movement, stomach pain and increase PT and APTT will be assessed. | from time of randomization till seven days
  o Adverse drug reactions related to ASX as increase bowel movement, stomach pain and increase PT and APTT will be assessed.
Length of hospital and ICU stay. | from time of randomization till seven days
  Length of hospital and ICU stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Elmatarya Teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Youssef FM, Ateyya H, Hanna Samy AE, Elmokadem EM. The anti-inflammatory and antioxidant effects of astaxanthin as an adjunctive therapy in community-acquired pneumonia: a randomized controlled trial. Front Pharmacol. 2025 Aug 7;16:1621308. doi: 10.3389/fphar.2025.1621308. eCollection 2025. PMID 40852606